CLINICAL TRIAL: NCT03756857
Title: Comparison of IVF Success Rates Between Different Embryo Transfer Techniques: Afterload Technique and Trial Followed by Transfer Technique
Brief Title: Does the Embryo Transfer Technique Affect the Success of in Vitro Fertilization?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Acibadem Kadiköy Hospital (Other)
Responsible Party: Principal Investigator, deniz usal, Medical Doctor, Acibadem Kadiköy Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AcibademKD
Record Dates: First submitted 2018-11-27; First posted 2018-11-28 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Infertility; Assisted Reproductive Technology; IVF
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: Prospective, open, randomized, parallel, two-arm trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Afterload transfer (Experimental): First, an empty catheter passes to the level of the lower uterine segment under ultrasound guidance to a point where the inner catheter enters the endometrial cavity. The inner sheath is removed slowly, leaving the outer sheath just beyond the internal os. After verifying the catheter's position on the TA ultrasound scan, the physician gives the signal to the embryologist to start the embryo loading. The embryologist brings the loaded inner catheter and inserts it into the outer sheath, which is maintained in its position by the physician.
  Interventions: Procedure: Afterload Transfer
- Trial Followed by Transfer (Experimental): First a trial transfer is performed using both the inner catheter and outer sheath connected together in standard configuration, just before the actual embryo transfer. It is passed up to and just through the the internal os. When it appears that the actual transfer will be possible without great difficulty ,the trial catheter is withdrawn. An embryo transfer catheter is loaded and the actual transfer is performed
  Interventions: Procedure: Trial followed by transfer

INTERVENTIONS:
Procedure: Afterload Transfer — Embryo transfer is done by using "afterload transfer" method
  Arms: Afterload transfer
Procedure: Trial followed by transfer — Embryo transfer is done by using "afterload transfer" method
  Arms: Trial Followed by Transfer

SUMMARY:
Prospective, open, randomized, parallel, two-arm trial to compare the clinical pregnancy rate between most commonly used two embryo transfer techniques: trial followed by transfer technique and afterloading technique

DETAILED DESCRIPTION:
Eligible patients will be informed about the possibility of participating in the clinical trial in the beginning of treatment and on the day ET, a signed consent form will be collected from those recipients who confirmed their participation. These patients will be randomized immediately before the ET procedure by sequentially numbered, opaque, sealed envelopes

ELIGIBILITY:
Inclusion Criteria:

1. Patient has given written informed consent
2. BMI 18-30 kg/m2
3. < 2 previous failed IVF trials
4. At least two good quality embryos on the day of transfer

Exclusion Criteria:

1. Congenital uterine anomaly
2. Untreated endometrial polyp or fibroid distorting uterine cavity
3. Presence of hydrosalpinx 4.2 or more prior IVF trial failure

5.Moderate to severe endometriosis 6.Recurrent pregnancy loss history

Ages: 20 Years to 37 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 200 (Estimated)
Dates: Start 2019-01-21 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
clinical pregnancy rate | 5-6 weeks after embryo transfer
  the presence of gestational sac on ultrasound

SECONDARY OUTCOMES:
implantation rate | 3-4 weeks after embryo transfer
  the number of gestational sacs divided by the number of embryos transferred

CONTACTS AND LOCATIONS:
Locations (1):
- Acibadem Altunizade Hospital, Unit of ART, Istanbul, Turkey (Türkiye)